CLINICAL TRIAL: NCT01462474
Title: Phase I Study of Concurrent Chemoradiotherapy With Famitinib for Patients With Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Concurrent Chemoradiotherapy With Famitinib for Patients With Locally Advanced Nasopharyngeal Carcinoma
Acronym: FMTN-I-LNPC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMTN-I-LNPC
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2011-11

CONDITIONS: Locally Advanced Nasopharyngeal Carcinoma
Keywords: Concurrent Chemoradiotherapy
MeSH Terms: interventions — famitinib; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug: Famitinib (Experimental)
  Interventions: Drug: Famitinib; Drug: Cisplatin; Radiation: radiation（IMRT）

INTERVENTIONS:
Drug: Famitinib — Either at 12.5 mg, 16.5 mg、20 mg or 25 mg qd p.o., 2 weeks before concurrent chemoradiotherapy and D1-D49, exception D1, D22, and D43.
Drug: Cisplatin — 100 mg/m2, D1, D22, and D43(q3w)
Radiation: radiation（IMRT） — IMRT (Intensity-Modulated Radiation Therapy). Radiation is delivered to GTV at 70 Gy in 32-33 fractions, CTV1 at 60 Gy in 32-33 fractions and CTV2 at 54 Gy in 32-33 fractions

SUMMARY:
RATIONALE: Famitinib is a tyrosin-inhibitor agent targeting at c-Kit, VEGFR2, PDGFR, VEGFR3, Flt1 and Flt3. Phase I study of mono famitinib has shown that the drug's toxicity is manageable.

PURPOSE: This phase I trial is studying the safety and tolerance of concurrent chemoradiotherapy with famitinib for patients with locally advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed nasopharyngeal differentiation or undifferentiation carcinoma, WHO II or III
* Newly diagnosed T3-4N1（exception metastatic uni or bil retropharyngeal lymph nodes N1） or any TN2-3(7th UICC/AJCC) locally advanced nasopharyngeal carcinoma
* 18-65 years of age
* ECOG performance status of 0 or 1
* Life expectancy of more than 6 months
* At least one measurable lesion :MRI scan larger than 10 mm in diameter, malignant lymph nodes larger than 10 mm in short axis
* Female: All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 6 months after the last dose of test article. Child bearing potential, a negative urine or serum pregnancy test result before initiating Famitinib. Male: All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 6 months after the last dose of test article.
* Signed and dated informed consent. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

* Before or at the same time any second malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Any factors that influence the usage of oral administration
* Known Spinal Cord compression or diseases of brain or pia mater by CT /MRI Screening
* Imageology shows that tumor lesion less than 5 mm to great vessels(internal carotid and jugular vein)
* Hemoglobin < 90g/L, platelets < 100×10^9/L, neutrophils < 2×10^9/L, total bilirubin ≥ 1.25×the upper limit of normal(ULN), ALT\AST ≥ 1.5x ULN), serum creatine > 1x ULN, creatinine clearance rate < 60ml/min, Cholesterol > 7.75 mmol/L and triglyceride > 3 mmol/L, LVEF: < LLN
* Hypertensive( more than 140/90 mmHg ), more than class I (NCI CTCAE 3.0 ) myocardial ischemia, arrhythmia(including QTcF:male ≥ 450 ms, female ≥470 ms), or cardiac insufficiency
* URT: urine protein ≥ ++ and > 1.0 g of 24 h
* Long-term untreated wounds or fractures
* PT, APTT, TT, Fbg abnormal, having hemorrhagic tendency (eg. active peptic ulcer disease) or receiving the therapy of thrombolysis or anticoagulation
* Before the first treatment occurs artery / venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism, etc
* Preexisting thyroid dysfunction, even using medical therapy, thyroid function cannot maintain in the normal range
* Abuse of Psychiatric drugs or dysphrenia
* Subject of Viral hepatitis type B or type C
* Subject of immunodeficiency: HIV positive, or other acquired immunodeficiency, congenital immunodeficiency, or organ transplantation
* With drug CYP3A4 inhibitor, inducer, or substrate
* Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-10; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) | 3 weeks
  To evaluate the DLT and MTD in patients with Concurrent Chemoradiotherapy With Famitinib

SECONDARY OUTCOMES:
ORR (Objective Response Rate) | 12 weeks after treatment
OS(Overall Survival) | 2 years and 3 years
DFMR(Distant Free Metastases Rate) | 2 years and 3 years
DFSR(Disease Free Survival Rate) | 2 years and 3 years
LFRSR(Local Free Recurrence Survival Rate) | 2 years and 3 years
Quantitative evaluation of the blood perfusion of the metastatic cervical lymph nodes by dynamic contrast-enhanced ultrasonography after a loading dose of famitinib for 14 days | 2 weeks
To identify the tumor's molecular profiles in patients with NPCs | 2 years
To measure the changes of serum c-Kit，VEGF，Filt，KDR，and PDGFR | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Cancer Center, Sun Yet-sen University, Guangzhou, Guangdong, China